CLINICAL TRIAL: NCT01875510
Title: The Effect of Fish-oil Lipid Emulsions on Neonatal Cholestasis and Retinopathy of Prematurity
Brief Title: The Influence of Fish-oil Lipid Emulsions on Neonatal Morbidities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Serdar Beken, M.D., Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B.10.4.İSM.4.06.68.49/144
Record Dates: First submitted 2013-05-31; First posted 2013-06-11 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Retinopathy of Prematurity; Neonatal Cholestasis
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — SMOFlipid; Soybean Oil; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish-oil emulsions (Active Comparator): Fish-oil emulsions:Preterm infants will receive a fish-oil emulsion administered from the first day of life 1gr/kg, second day 2gr/kg and third day and after 3 gr/kg.
  Interventions: Dietary Supplement: Fish-oil emulsions; Dietary Supplement: soybean-oil emulsion
- soybean-oil emulsion (Placebo Comparator): Preterm infants will receive a soybean-oil emulsion administered from the first day of life 1gr/kg, second day 2gr/kg and the third day and after 3gr/kg
  Interventions: Dietary Supplement: Fish-oil emulsions; Dietary Supplement: soybean-oil emulsion

INTERVENTIONS:
Dietary Supplement: Fish-oil emulsions — Fish -oil emulsions:
  Preterm infants will receive a fish-oil emulsion administered from the first day of life 1gr/kg, second day 2gr/kg and third day and after 3 gr/kg.
  Other Names: Smoflipid
Dietary Supplement: soybean-oil emulsion — soybean-oil emulsion
  Other Names: Intralipid

SUMMARY:
Docosahexaenoic acid (DHA) has been shown to be particularly important for fetal and neonatal development. Infants born prematurely are at special risk for DHA insufficiency. The source of DHA after birth for preterm babies who are not fed full enterally, are mostly fat emulsions as the component of total parenteral nutrition solutions which usually do not contain DHA. The aim of this study is to investigate if the fish oil emulsion-administered from the first day of life and during parenteral nutrition-prevents infants from cholestasis and retinopathy of prematurity.

DETAILED DESCRIPTION:
During the study period, preterm infants admitted to NICU were included. Infants who weighed <1500 gr and delivered prematurely before the 32nd week of gestation were eligible for the study. Infants with major congenital anomalies, congenital infections and inborn metabolic errors were excluded from the study.

Group 1: Fish-oil emulsion (20% SMOFLipid: soybean oil 60 g/dL, MCT 60 g/dL, olive oil 50 g/dL, fish oil 30 g/dL, egg phospholipids 12 g/dL, glycerol 25 g/dL, vitamin E 200 mg α-TE/L) Group 2: Soybean oil emulsion (20% Intralipid: soybean oil 200 g/dL, egg phospholipids 12 g/dL, glycerol 22,5 g/dL, vitamin E 57 mg α-TE/L).

ELIGIBILITY:
Inclusion Criteria:

* Infants below 32 gestational age and requiring parenteral nutrition

Exclusion Criteria:

* Infants with congenital anomalies, infants above 32 gestational age

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Beken, Principal Investigator — Dr. Sami Ulus Children's Hospital
Locations (1):
- Dr. Sami Ulus Childrens Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Pawlik D, Lauterbach R, Turyk E. Fish-oil fat emulsion supplementation may reduce the risk of severe retinopathy in VLBW infants. Pediatrics. 2011 Feb;127(2):223-8. doi: 10.1542/peds.2010-2427. Epub 2011 Jan 3. PMID 21199856

RESULTS

PARTICIPANT FLOW:
Groups:
- Fish-oil Emulsions: Preterm infants will receive a fish-oil emulsion administered from the first day of life 1gr/kg, second day 2gr/kg and third day and after 3 gr/kg.
Period: Overall Study
Arm/Group | Fish-oil Emulsions | Soybean-oil Emulsion
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish-oil Emulsions | Soybean-oil Emulsion | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 40 | 80
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks]
  gestational age | 30 (2) | 30 (3) | 30 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  Turkey | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Retinopathy of Prematurity
Description: The number of Participants with Retinopathy of Prematurity will be defined.
Time Frame: Corrected age 32 weeks or postnatal 28th day
Measure: Number; unit: participants
Arm/Group | Fish-oil Emulsions | Soybean-oil Emulsion
Number analyzed (Participants) | 40 | 40
participants | 2 | 13

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fish-oil Emulsions | Soybean-oil Emulsion
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
The limitation of our study is that participants are mostly above 1000 grams. It was a single center study and DHA levels were not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes